CLINICAL TRIAL: NCT06318676
Title: A Phase 1, Multi-center, Open-label, Single-dose Study to Assess the Pharmacokinetics of Mezigdomide (BMS-986348, CC-92480) in Adult Participants With Normal Renal Function, Severe Renal Impairment, and End-stage Renal Disease
Brief Title: A Study to Evaluate the Drug Levels of Mezigdomide in Adult Participants With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA057-1009
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Renal Impairment
Keywords: Chronic Kidney Disease; End Stage Renal Disease; Dialysis; Hemodialysis; Mezigdomide; Pharmacokinetics; Healthy
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A: Participants with severe renal impairment (Experimental)
  Interventions: Drug: Mezigdomide
- Group B: Participants with End Stage Renal Disease (Experimental)
  Interventions: Drug: Mezigdomide
- Group C: Participants with normal renal function (Experimental)
  Interventions: Drug: Mezigdomide

INTERVENTIONS:
Drug: Mezigdomide — Specified dose on specified days
  Other Names: BMS-986348; CC-92480

SUMMARY:
The purpose of this study is to evaluate the drug levels of mezigdomide in participants with renal impairment.

ELIGIBILITY:
Inclusion Criteria

* Participants must have a body mass index (BMI) of ≥ 18.0 kg/m2 to ≤ 40.0 kg/m2 inclusive at screening.
* Participants must have a body weight ≥ 50 kg at screening.
* Participants must be afebrile (febrile is defined as ≥ 38°C or 100.4°F) at screening, check in, and predose.

Exclusion Criteria

* Participants must not have any history of chronic pruritus or dermatologic syndromes that may be confounded with reactions to mezigdomide.
* Participants must not have any history of malignancy of any type other than in situ cervical cancer or surgically excised non-melanomatous skin cancers.
* Participants with an inability to tolerate oral medication.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to 24 days
Area under the plasma concentration-time curve (AUC) | Up to 24 days
Area under the plasma concentration-time curve from time 0 to time of last quantifiable concentration (AUC(0-T)) | Up to 24 days

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 54 days
Number of participants with serious adverse events (SAEs) | Up to 54 days
Number of participants with physical examination findings | Up to 24 days
Number of participants with vital sign abnormalities | Up to 24 days
Number of participants with 12-lead electrocardiogram (ECG) findings | Up to 24 days
Maximum observed concentration (Cmax) | Up to 24 days
Time of maximum observed concentration (Tmax) | Up to 24 days
Area under the plasma concentration-time curve (AUC) | Up to 24 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - PANAX, Miami Lakes, Florida
  - Omega Research Group - Orlando, Orlando, Florida
  - Orlando Clinical Research Center OCRC, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com